CLINICAL TRIAL: NCT04714060
Title: A Randomized, Single-blind, Dose-selected Phase II Trial to Evaluate the Safety and Efficacy of UB-621 in Adults With Recurrent Genital HSV-2 Infection
Brief Title: UB-621, a New Type of Anti-herpes Simplex Virus (HSV) Monoclonal Antibody for the Use in the Treatment of Adult Recurrent HSV-2 Infections of the Genitals
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: UBP Greater China (Shanghai) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UBP-A228-HSV
Record Dates: First submitted 2021-01-15; First posted 2021-01-19 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Recurrent Genital Herpes
MeSH Terms: conditions — Herpes Genitalis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cohort 1 (Experimental): 2.5 mg/kg UB-621 group
  Interventions: Biological: UB-621
- cohort 2 (Experimental): 5 mg/kg UB-621 group
  Interventions: Biological: UB-621

INTERVENTIONS:
Biological: UB-621 — mAb by SC administration

SUMMARY:
A randomized, single-blind, dose-selected phase II trial to evaluate the safety, efficacy and PK of UB-621 in adults with recurrent genital HSV-2 infection

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age inclusive.
* Subject must be HSV-2 seropositive
* Subjects have a history of recurrent genital herpes in the past year
* Subjects have a negative result on the HIV Ab/Ag assay
* Subjects must agree to use contraception during study participation
* Subjects must be willing to collect a swab each day from their genital area (non-lesional as well as lesional, if appropriate) during the swabbing periods, which are 8 weeks period after the administration of study drug.
* Subject must be willing to go back to the hospital within 72 hours after the new lesions are shown in the anal and genital area.
* Subject must be willing to observe the syndromes around the anal and genital area during study period, to evaluate the lesions according to the HSV lesion score, and to record in the patient dairy
* Female subjects must have a negative serum β-HCG at Screening and a negative urine pregnancy test prior to study drug administration.

Exclusion Criteria:

* Serious medical conditions, including poorly controlled diabetes, significant autoimmune diseases, co-existing sexually transmitted disease presentation (except HSV) in the anogenital area, etc. that may interfere with the assessment of the efficacy of UB-621.
* History or current evidence of malignancy except for a localized non-melanoma skin cancer
* Known immunosuppression
* Exposure to HSV vaccine
* Medical history of macular or maculopapular skin reactions to antibody (ie, as evidenced by IgG or plasma administration)
* Any other conditions that in the judgment of the Investigator would preclude successful completion of the clinical study
* Treatment with systemic steroids or other immunomodulating agents within 30 days prior to Screening or planned treatment with systemic steroids or immunomodulators during the study period.
* Renal impairment and/or hepatic impairment
* ECG abnormalities of clinical relevance or cardiovascular conditions
* Abnormal blood tests according to "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trial "in the Guidance for Industry, 2007:

  1. albumin<3 g/dl
  2. ALP>2.5*ULN
  3. ALT>2.5*ULN
  4. AST>2.5*ULN
  5. Bilirubin>1.5*ULN
  6. CPK>1.5*ULN
  7. rGGT>2.5*ULN
  8. Hemoglobin: female<11 g/dl; male<12.5 g/dl
  9. platelet<125*10E3/ul
  10. WBC<2.5*10E3/ul or
  11. ANC<1.5*10E3/ul

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with episodes before and after UB-621 treatment (self-comparison) | 16 weeks
  Proportion of subjects with episodes is calculated as the number of subjects with episodes divided by the number of total subjects. Primary endpoint is the self-comparison of proportion of subjects with episodes before and after UB-621 treatment.

SECONDARY OUTCOMES:
Lesion rate | 16 weeks
  Lesion rate is calculated as the number of days with lesion divided by the number of study days.
Duration of recurrent lesions | 16 weeks
  Duration of recurrent lesions is calculated as consecutive days with lesions of HSV score 2-7.
Recurrence rate | 16 weeks
  Recurrence rate is defined as number of recurrences divided by the total number of study days.
Time to first recurrence of lesion | 16 weeks
  Time to first recurrence of lesion as reported by patient and verified by investigator.

OTHER OUTCOMES:
HSV-2 shedding rate. | 8 weeks
  Viral shedding rate is defined as the number of positive anogenital swabs divided by total number of swabs.
Clinical and Subclinical HSV-2 Shedding Rates | 8 weeks
  Daily record of subject self-assessment of genital lesions in subject diary in addition to anogenital swabs collected daily from subjects during the follow-up periods will be used to evaluate the clinical (lesional) and subclinical (non-lesional) HSV-2 shedding rates.
Rate of HSV-2 Shedding Episodes | 8 weeks
  The rate of HSV-2 shedding episodes is the number of onsets of shedding episodes divided by the total number of days with swabs collected. Shedding episodes are defined as consecutive HSV-2 positive swab results including no more than 1 consecutive negative result or missed swab. The episodes are preceded and followed by 2 consecutive negative swab results.
HSV-2 viral load | 8 weeks
  Anogenital swab samples collected from subjects during follow-up period will be used to quantify HSV-2 DNA copies.

IPD SHARING:
Plan to Share IPD: No